CLINICAL TRIAL: NCT03107364
Title: Association Between Trend in Length of Stay and Risk of Readmission at Hospital After Surgery
Brief Title: Trend in Hospital Lengths of Stay and Readmissions
Acronym: ELIPSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0036
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Trend in Hospital Lengths of Stay and Readmissions
MeSH Terms: interventions — Length of Stay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal surgery: Patient who underwent elective colorectal surgery
  Interventions: Other: Hospital stay
- Hip fracture: Patient who underwent urgent surgical procedure for hip fracture
  Interventions: Other: Hospital stay

INTERVENTIONS:
Other: Hospital stay — Collection of hospital lengths of stay and readmissions

SUMMARY:
Medical and surgical innovations have allowed to shorter length of hospital stay (LOS). We assume that hospitals with uncontrolled reduction in LOS may expose patients to unsafe care. At the institutional level, a dynamic analysis of LOS evolution over time could clarify the existence of a link with the risk of readmission.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent elective colorectal surgery or urgent surgical procedure for hip fracture in French public and private hospitals from January 2014 to December 2016

Exclusion Criteria:

* Age < 18 years old
* Death during the index stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated for colorectal disease or hip fracture
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Unplanned hospital readmission with death, intensive care, or reoperation | 30 days
  Number of unplanned hospital readmission with death, intensive care, or reoperation within 30 days of surgical procedure

SECONDARY OUTCOMES:
Unplanned hospital readmission with death, intensive care, or reoperation | 3 months
  Number of unplanned hospital readmission with death, intensive care, or reoperation within 3 months of surgical procedure
Unplanned hospital readmission with death, intensive care, or reoperation | 6 months
  Number of unplanned hospital readmission with death, intensive care, or reoperation within 6 months of surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Antoine DUCLOS, MD, PhD, Principal Investigator — Pôle Information Médicale Evaluation Recherche des Hospices Civils de Lyon
Locations (1):
- Pôle Information Médicale Evaluation Recherche des Hospices Civils de Lyon, Lyon, France